CLINICAL TRIAL: NCT01362283
Title: A Multi-center, Observational, Cross-sectional Study to Evaluate CVD Risk Factors in Korean Hypertensive Patients
Brief Title: Epidemiologic Study to Evaluate the Proportion of Cardiovascular Disease Risk Factors in Korean Hypertensive Patients
Acronym: WONDeR
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114619
Record Dates: First submitted 2011-05-05; First posted 2011-05-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertension: Subject who meet eligible criteria
  Interventions: Other: Blood Sampling

INTERVENTIONS:
Other: Blood Sampling — Blood sampling for Fasting Plasma Glucose, Hemoglobin A1C, Cholesterols, Blood Urea Nitrogen, Creatinine
  Other Names: Blood sampling for cardiovascular disease risk

SUMMARY:
The purpose of this study is investigating the proportion of Cardiovascular disease risk factors of hypertensive patients.

DETAILED DESCRIPTION:
Primary endpoint: To evaluate the Proportion of patients with Cardiovascular disease high risk factors

Secondary endpoint: To evaluate the Proportion of patients with Cardiovascular disease risk factors, To evaluate the Proportion of patients with Cardiovascular disease, To evaluate Target blood pressure achievement rate according to the proportion of Cardiovascular disease risks

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertensive patient no less than 18 yeas old
* Patient who gave informed consent form

Exclusion Criteria:

* Patient was diagnosed as secondary hypertension
* Patient who have white-coat hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korea, Diagnosed hypertensive patient
Sampling Method: Probability Sample
Enrollment: 3109 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with cardiovascular disease high risk factors | 6years, average duration of hypertension
  Between patients with essential hypertension

SECONDARY OUTCOMES:
Proportion of patients with Cardiovascular disease risk factors | 6years, average duration of hypertension
  Between patients with essential hypertension
Proportion of patients with Cardiovascular disease | 6years, average duration of hypertension
  Between patients with essential hypertension
Target Blood Pressure achievement rate according to the proportion of Cardiovascular disease risks | 6years, average duration of hypertension
  Between patients with essential hypertension

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline